CLINICAL TRIAL: NCT02708316
Title: The Gut Metagenome Research of Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Rehabilitation Hospital of Bao Ji City (Unknown); Center Hospital of Xian Yang City (Unknown); Mental Health Center of Wei Nan City (Unknown)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRS-2015-009
Record Dates: First submitted 2016-03-03; First posted 2016-03-15 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool samples retained for sequencing faecal metagenome

GROUPS / COHORTS (2):
- schizophrenia group: schizophrenia patients in the group
  Interventions: Genetic: sequencing faecal metagenome
- control group: healthy population
  Interventions: Genetic: sequencing faecal metagenome

INTERVENTIONS:
Genetic: sequencing faecal metagenome — sequencing faecal metagenome is not the intervention measure.It is the observational method for investigators to detect the component of faecal microorganism.

SUMMARY:
Research already found that patients with autistic spectrum disorders lack of Prevotella intestinal type, then schizophrenia patients may also show the specific intestinal type, so investigators want to detect the gut metagenome of schizophrenia patients by high-throughput DNA sequencing to find specific intestinal type, so as to achieve the purpose of schizophrenia diagnosis. According to the detection of inflammatory factors in the blood, nerve growth factor in the cerebrospinal fluid, to find the mechanism of the gut-microbes-brain axis. Furthermore, investigators want to identify intestinal strains involved in weight gain and metabolic disorders such as blood glucose and lipids induced by antipsychotic drugs.

DETAILED DESCRIPTION:
A prospective observational study will be conducted and cases will be recruited by multi-center cooperation. Investigators plan to collect 100 schizophrenic patients as case group, 100 healthy people as control group. Investigators will observe schizophrenia patients who use the single drug of risperidone in the treatment and follow up the patients on day 1, the third week, the third month, the sixth month and the first year. In addition, the other two groups of patients with schizophrenia will be included, one with olanzapine and the other with aripiprazole. There are three objectives:

1. Compare healthy population with schizophrenia patients in the difference of gut metagenome and inflammatory factors in the blood, stool samples aimed at detecting the difference of composition of intestinal microorganism;
2. Observe the change of intestinal microorganism, inflammatory factors, γ-aminobutyric acid of schizophrenic patients who received risperidone treatment according to the blood, stool samples, cerebrospinal fluid during the follow-up period.
3. Study the difference of intestinal flora composition between schizophrenia patients with metabolic disorder and schizophrenia patients without metabolic disorder after olanzapine or aripiprazole treatment and discuss the relationship between intestinal flora composition and metabolic disorder.

ELIGIBILITY:
Inclusion Criteria:

* The first episode or recurrent acute-exacerbation schizophrenia patients who correspond to the Diagnostic and Statistical Manual of Mental Disorders-Ⅵ (DSM-Ⅵ) diagnostic criteria.
* Between 18 and 45 years old (including 18 and 45 years old, male or female).
* Patients never accepted full range of psychotropic drugs before admission(taking psychotropic drug less than 5 days before admission)
* the duration of recurrent patients is less than 5 years
* the period of taking psychiatric drug before admission is no more than 2 weeks.
* didn't use of antibiotics within consecutive 3 days in recent 3 months.
* meet the indications of a single antipsychotic risperidone treatment.
* All the patients must have a good family support and comply with the requirements and signed informed consent
* The PANSS score is greater than 60 or equal to 60.
* BMI is greater than or equal 17.5 and less than or equal to 30.

Exclusion Criteria:

* Patients have severe unstable cardiovascular disease, liver disease, kidney disease, blood disease and endocrine disease or history.
* Patients have the history of systematic disease or history of malignant tumor or relevant complications.
* Patients have the activity of gastrointestinal diseases.
* Patients have organic brain disease or complications and mental retardation.
* According to the DSM-Ⅵ diagnostic criteria , patients have drug abuse or drug dependence and incomplete remission.
* glutamic-oxalacetic transaminase (AST) or glutamic-pyruvic transaminase (ALT) is 2 times higher than the normal limit.
* Renal dysfunction, creatinine is higher than the upper limit of normal value.
* The women in pregnancy or lactation now, and may be in pregnant during the study period.
* Patients are allergic to risperidone.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The cases included the first episode or recurrent acute-exacerbation schizophrenia patients who correspond to the DSM-Ⅵ diagnostic criteria. The healthy population is matched with cases based on gender, age, nationality, smoking, diet, education and socioeconomic status.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-04; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
species-level molecular operational taxonomic units | at the beginning
  The composition of the gut microbe was evaluated by sequencing faecal metagenome. The specific measures representing the above characteristics of gut microbe contain species-level molecular operational taxonomic units.
species-level molecular operational taxonomic units | the third month
  The composition of the gut microbe was evaluated by sequencing faecal metagenome. The specific measures representing the above characteristics of gut microbe contain species-level molecular operational taxonomic units.

SECONDARY OUTCOMES:
concentration of inflammatory factors | at the beginning
  concentration of inflammatory factors including interleukin-1(IL-1),interleukin-10(IL-10),interleukin-2 (IL-2),interleukin-6 (IL-6),tumor necrosis factor (TNF), the measure unit is U/mL
concentration of inflammatory factors | the third week
  concentration of inflammatory factors including IL-1,IL-10,IL-2,IL-6,TNF, the measure unit is U/mL
concentration of inflammatory factors | the third month
  concentration of inflammatory factors including IL-1,IL-10,IL-2,IL-6,TNF, the measure unit is U/mL
concentration of inflammatory factors | the sixth month
  concentration of inflammatory factors including IL-1,IL-10,IL-2,IL-6,TNF, the measure unit is U/mL
concentration of inflammatory factors | one year
  concentration of inflammatory factors including IL-1,IL-10,IL-2,IL-6,TNF, the measure unit is U/mL
concentration of γ-aminobutyric acid | at the beginning
  γ-aminobutyric acid was measured by high efficiency liquid chromatography in cerebrospinal fluid, the measure unit is mg/kg
concentration of γ-aminobutyric acid | the sixth month
  γ-aminobutyric acid was measured by high efficiency liquid chromatography in cerebrospinal fluid, the measure unit is mg/kg
gene profiles | at the beginning
  The composition of the gut microbe was evaluated by sequencing faecal metagenome. The specific measures representing the above characteristics of gut microbe contain gene profiles.
gene profiles | the third month
  The composition of the gut microbe was evaluated by sequencing faecal metagenome. The specific measures representing the above characteristics of gut microbe contain gene profiles.
metagenomic linkage groups | at the beginning
  The composition of the gut microbe was evaluated by sequencing faecal metagenome. The specific measures representing the above characteristics of gut microbe contain metagenomic linkage groups.
metagenomic linkage groups | the third month
  The composition of the gut microbe was evaluated by sequencing faecal metagenome. The specific measures representing the above characteristics of gut microbe contain metagenomic linkage groups.
Encyclopedia of Genes and Genomes (KEGG) ortholog | at the beginning
  The composition of the gut microbe was evaluated by sequencing faecal metagenome. The specific measures representing the above characteristics of gut microbe contain Encyclopedia of Genes and Genomes (KEGG) ortholog.
Encyclopedia of Genes and Genomes (KEGG) ortholog | the third month
  The composition of the gut microbe was evaluated by sequencing faecal metagenome. The specific measures representing the above characteristics of gut microbe contain Encyclopedia of Genes and Genomes (KEGG) ortholog.
module and pathway profiles of faecal microbiota | at the beginning
  The composition of the gut microbe was evaluated by sequencing faecal metagenome. The specific measures representing the above characteristics of gut microbe contain module and pathway profiles of faecal microbiota.
module and pathway profiles of faecal microbiota | the third month
  The composition of the gut microbe was evaluated by sequencing faecal metagenome. The specific measures representing the above characteristics of gut microbe contain module and pathway profiles of faecal microbiota.

CONTACTS AND LOCATIONS:
Overall Officials: Xiancang Ma, MD,PHD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China